CLINICAL TRIAL: NCT04808011
Title: A Single Arm, Prospective, Open Label, Cross-Over, Multi-Center Study to Evaluate the Safety, Feasability and Usability of the Intelligent Dialysis Assistant (IDA)
Brief Title: A Single Arm, Multi-Center Study To Evaluate The Intelligent Dialysis Assistant (IDA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: liberDi Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP-028-20
Record Dates: First submitted 2021-03-01; First posted 2021-03-19 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Chronic Kidney Disease Stage 5
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The subjects will undergo a single peritoneal dialysis exchange procedure at the PD clinic, under the supervision of the medical staff and instructed about its operation. Further exchanges will be performed by the subjects themselves at home.
  The study includes two cohorts and two phases: in the first phase (phase I), 20 subjects will be recruited as Cohort 1 to undergo a single exchange in the medical center using the IDA. Following the completion of recruitment of all 20 subjects and the performance of the single on site exchange, the Sponsor will perform an interim analysis of the results for safety and initial feasibility, followed by submission of the results to the MoH and approval of the second phase (phase II).
  Subjects will be treated with their routine dialysis device for 14 days, followed by a treatment with the IDA for a period of 30 days, and then an additional period of 14 days of treatment with their routine dialysis device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Each subjects will be treated with his prescribed dialysis device for 14 days, followed by a treatment period of 30 days with the investigational IDA system, and concluding with additional 14 days of treatment with the prescribed dialysis device.
  Interventions: Device: Intelligent Dialysis Assistant (IDA)

INTERVENTIONS:
Device: Intelligent Dialysis Assistant (IDA) — The IDA is intended for home dialysis for subjects who are stage 5 kidney diease patients and who perform Peritoneal Dialysis. The system is used deveral times a day for approximately 20 minutes for each cycle. During the interventional period, subjects will use only the investigational IDA system for their in/out exchanges.

SUMMARY:
This is a multi-center, open label, cross-over clinical study. A total of 18 subjects will be enrolled to use the IDA for every peritoneal dialysis exchange for 14 days. To participate in the study, the subjects must have current CKD5 and have been treated with PD for at least 3 months. The subjects will undergo a single peritoneal dialysis exchange procedure at the PD clinic, under supervision of the medical staff and instructed about its operation. Further exchanges will be performed by the subjects themselves at home.

The study includes three periods:

1. First period (Observational): 14-day Observational Period. Eligible subjects who sign informed consent will continue with their regular CAPD treatment while performing measurement and recording of dialysate in/out time.
2. Second period (Interventional): 14-day interventional period, where subjects will perform dialysis exchanges using the IDA according to the below visit schedule.
3. Third period (Follow up): 14-day follow up period, during which the study staff will call the subject once weekly to inquire about device-related SAEs and any changes to concomitant medications.

DETAILED DESCRIPTION:
This is a multi-center, open label, cross-over clinical study. A total of 20 subjects will be enrolled to use the IDA for every peritoneal dialysis exchange for 14 days. To participate in the study, the subjects must have current CKD5 and have been treated with PD for at least 3 months. The subjects will undergo a single peritoneal dialysis exchange procedure at the PD clinic, under supervision of the medical staff and instructed about its operation. Further exchanges will be performed by the subjects themselves at home.

The study includes two cohorts and two phases: in the first phase (phase I), 20 subjects will be recruited as Cohort 1 to undergo a single exchange in the medical center using the IDA. Following the completion of recruitment of all 20 subjects and the performance of the single on site exchange, the Sponsor will perform an interim analysis of the results for safety and initial feasibility, followed by submission of the results to the MoH and approval of the second phase (phase II). The expected timeframe between phase I and phase II is up to 4 weeks. An additional cohort, Cohort 2, will be added to Phase I, which will include additional ten (10) subjects. These subjects will undergo the same procedure at the dialysis clinic, with the addition of blood sampling for CBC and Chemistry two (2) hours ±30 minutes after the procedure. A total of 20 subjects from either cohort, meeting the inclusion and exclusion criteria of Cohort 1, will continue to complete the second phase of the study (Phase II).

Phase II of the study includes three periods:

First period (Observational): 14-day Observational Period. Eligible subjects who sign informed consent will continue with their regular CAPD treatment while performing measurement and recording of dialysate in/out time.

Second period (Interventional): 14-day interventional period, where subjects will perform dialysis exchanges using the IDA according to the below visit schedule.

Third period (Follow up): 14-day follow up period, during which the study staff will call the subject once weekly to inquire about device-related SAEs and any changes to concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CKD stage 5 treated by continuous ambulatory peritoneal dialysis (CAPD)
* Male or female, Age >18 years
* Mental ability to understand study procedures and provide an informed consent
* More than 3 months on PD (Peritoneal Dialysis)
* At least 3 daily exchanges
* Self-treated subject
* Stable PD prescription for the last month

Exclusion Criteria:

* Need of cycler (APD, Automated Peritoneal Dialysis)
* Known mechanical problem (drainage, fill) during the last month prior to enrollment
* Pregnant or breastfeeding women
* subject who is unwilling or unable to comply with study procedures
* Known Peritonitis or other catheter associated infections during the last 3 months prior to enrollment
* Known Congestive heart failure stage III- IV
* Non-elective hospitalization during the last 3 months prior to enrollment
* Any other medical or mental condition, that at the investigator's discretion may prevent the subject from participating in the study
* Participation in any other clinical study within 4 weeks prior to enrollment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Device-Related Serious Adverse Event Incidence | 14 days
  Incidence of device-related SAEs throughout the active investigational phase (14 days).
AE during on site exchange | 1 day
  Incidence of device-related adverse events during the on-site exchange - phase I of the study.

SECONDARY OUTCOMES:
Procedure Time Length | 14 days
  Time length of the in/out PD exchange procedure.
Usability Questionnaire | 14 days
  completion of a Usability questionnaire, designed by the Sponsor, which reflects the physician's impression by the device usage. The questionnaire consists of 4 questions devided to "yes/no" sub-questions.
Device-Related Serious Adverse Events Incidence During Follow Up Period | 14 days
  Incidence of device-related SAEs during the additional 14-day follow up period
Renal Treatment Internal Questionnaire | 42 days
  Analysis of the subject's treatment feedback and effect on quality of life, provided to him/her by using the device. The questionnaire consists of 6 questions ranked from 1 (very dissatisfied) to 5 (very satisfied). The Total Score will be calculated for this questionnaire, with a range of 6-30. A score above 18 will be considered "satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Tansyochuk, MD, Principal Investigator — Carmel MC, Haifa
Locations (3):
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Carmel MC, Haifa
  - Meir Medical Center, Kfar Saba

IPD SHARING:
Plan to Share IPD: No